CLINICAL TRIAL: NCT03670134
Title: The Use of Volumetric Laser Endomicroscopy to Predict Recurrence of Barrett's Esophagus After Complete Eradication of Intestinal Metaplasia
Brief Title: Predict Recurrence of Barrett's Esophagus After Complete Eradication of Intestinal Metaplasia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The company that supported the technology (volumetric laser endomicroscopy) is no longer operational due to the pandemic.
Sponsor: Mayo Clinic (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other)
Responsible Party: Principal Investigator, Cadman Leggett, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-003333
Record Dates: First submitted 2018-08-30; First posted 2018-09-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Barrett Esophagus
Keywords: Laser Endomicroscopy; Intestinal Metaplasia
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Volumetric laser Endomicroscopy (VLE) (Experimental): Volumetric laser Endomicroscopy (VLE) is a second-generation optical coherence tomography platform that can image the human esophagus in cross-section at microscopic resolution this will performed by using the Nvision VLE Imaging System.
  Interventions: Device: The Nvision VLE Imaging System

INTERVENTIONS:
Device: The Nvision VLE Imaging System — Volumetric laser Endomicroscopy (VLE) will be performed by using the Nvision VLE Imaging System (Nine Point Medical, MA) consists of an imaging console, monitor and optical probe. The optical probe is centered by a balloon (diameter: 14 mm, 17 mm, 20 mm; length: 6 cm) that is deployed through a diagnostic gastroscope's instrument channel. Imaging is performed by automatic helical pullback of the probe from the distal to the proximal end of the balloon over 90 seconds.

SUMMARY:
Researchers are trying to see if the Nvision® Imaging System (VLE) can accurately determine the risk of recurrent Barrett's esophagus in patients with Barrett's esophagus which have been clear of disease.

DETAILED DESCRIPTION:
Patients with Barrett's Esophagus (BE) undergoing endoscopic therapy through our Barrett's Esophagus Unit will be approached for study enrollment. Patients with no endoscopic evidence of BE will be considered for the study. Surveillance biopsies will be obtained per standard clinical protocol and reviewed to confirm absence of intestinal metaplasia. Patients who have achieved complete eradication of intestinal metaplasia (CRIM) will be enrolled in the study and will undergo the Nvision® Imaging System (VLE). Patients enrolled in the study will undergo clinical follow-up consisting of surveillance endoscopy every 3 months for 1 year. Surveillance endoscopy intervals may be prolonged to every 6 months in the second year, and annually thereafter. At each follow-up visit, endoscopic data will be collected to determine if patients remain in CRIM or show evidence of recurrent disease. Patients will be followed for 1 year (endpoint 1) and 3 years (endpoint 2).

.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing an upper endoscopy with prior biopsy confirmed Barrett's Esophagus.
* Ability to provide written, informed consent
* No significant esophagitis (LA grade <B, C, and D)

Exclusion Criteria:

* Patients for whom use of the NvisionVLE device would be in conflict with the instruction for use.
* Prior esophageal or gastric surgical resection
* Significant esophageal stricture requiring dilatation
* Patients who require anti-coagulation for who biopsy would be contraindicated
* Patients who are known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Determine association between number of glandular structures measured with volumetric laser endomicroscopy and recurrence of Barrett's esophagus following endoscopic therapy | 1 year
  Measure the number of glandular structures observed with volumetric laser endomicroscopy in patients who remain free of Barrett's esophagus and in those with recurrent disease. Report the mean and standard-deviation of this metric and determine a statistical significant difference using the Student's t-test.
Determine association between distribution of glandular structures measured with volumetric laser endomicroscopy and recurrence of Barrett's esophagus following endoscopic therapy | 1 year
  Measure the distribution (gastric cardia versus esophagus) of glandular structures observed with volumetric laser endomicroscopy in patients who remain free of Barrett's esophagus and in those with recurrent disease. Report the mean and standard-deviation of this metric and determine a statistical significant difference using the Student's t-test.
Determine association between thickness of neosquamous epithelium measured with volumetric laser endomicroscopy and recurrence of Barrett's esophagus following endoscopic therapy | 1 year
  Measure the thickness of neosquamous epithelium (mm) with volumetric laser endomicroscopy in patients who remain free of Barrett's esophagus and in those with recurrent disease. Report the mean and standard-deviation of this metric and determine a statistical significant difference using the Student's t-test.

SECONDARY OUTCOMES:
Develop a volumetric laser endomicrosopy feature scoring index to stratify the risk of disease recurrence in patients with Barrett's esophagus following treatment | 3 years
  The proposed model will stratify patients into two categories (1) low risk of recurrence and (2) high risk of recurrence. Low risk of disease recurrence is defined by a rate of <5% per patient-year. High risk of disease recurrence is defined by a rate of >10% per patient year.

CONTACTS AND LOCATIONS:
Overall Officials: Cadman L Leggett, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials